CLINICAL TRIAL: NCT00545974
Title: A Prospective, Randomized, Multi-Center, Double-Blind, 26 Week, Placebo-Controlled Trial of Memantine (10mg BID) for the Frontal and Temporal Subtypes of Frontotemporal Dementia
Brief Title: Memantine (10mg BID) for the Frontal and Temporal Subtypes of Frontotemporal Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAM-53:memantineplacebo
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Frontal Lobe Dementia; Frontotemporal Lobe Dementia; Semantic Dementia
Keywords: Randomized; Double-Blind; Placebo-Controlled; memantine; Namenda; Frontotemporal Dementia; Semantic Dementia; FTD; SD; dementia; behavioral decline; cognitive decline
MeSH Terms: conditions — Frontotemporal Dementia; Dementia; Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Memantine 10mg BID
  Interventions: Drug: memantine
- 2 (Placebo Comparator): Placebo condition
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: memantine — memantine 10mg BID
  Arms: 1
Drug: Placebo pill — Placebo pill BID
  Arms: 2

SUMMARY:
The primary objective of the study is to determine whether memantine is effective in slowing the rate of behavioral decline in frontotemporal dementia.

The secondary objective of the study is to assess the safety and tolerability of long-term treatment with memantine in patients with frontotemporal dementia (FTD) or semantic dementia (SD). To determine whether memantine is effective in slowing the rate of cognitive decline in frontotemporal dementia. To evaluate whether memantine delays or decreases the emergence of parkinsonism in frontotemporal dementia.

The tertiary objective of the study is to determine whether treatment with memantine affects changes in weight

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial of memantine 10 mg twice daily versus placebo, at a ratio of 1:1, to receive active drug or placebo. Screening and enrollment is planned to last approximately one year. A Data and Safety Monitoring Board, consisting of a clinical pharmacist and 3 neurologists will review all AE reports approximately every 3 months after study initiation. The DSMB will notify the principal investigator, the study sponsor and the CHR if significant concerns are raised by their review of the AE data. An interim analysis of efficacy data will be conducted after 50% of the targeted enrollment population has completed 26 weeks of drug treatment.

Including screening and off-drug follow up, each subject will participate in the study for approximately 34 weeks.

The entire study is anticipated to last 86 weeks if enrollment is completed within one year of study initiation.

The targeted enrollment is 140.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet ALL of the following criteria to be considered for enrollment in this study:

1. Signed and dated written informed consent obtained from the subject and the subject's caregiver in accordance with local IRB regulations.
2. Must meet criteria Neary et al. criteria for frontotemporal dementia (FTD) or semantic dementia (SD)
3. Age: 40-80
4. CT or MRI of brain within 12 months consistent with a diagnosis of FTD or SD.
5. MMSE ≥ 15 at screening visit.
6. Judged by investigator to be able to comply with neuropsychological evaluation at baseline.
7. Must have reliable caregiver accompany subject to all study visits. Caregiver must read, understand and speak English fluently in order to ensure comprehension of informed consent form and informant-based assessments of subject. Caregiver must also have frequent contact with subject (at least 3 times per week for one hour) and be willing to monitor study medication compliance and the subject's health and concomitant medications throughout the study.
8. In the opinion of the investigator, the patient and the caregiver will be compliant with the protocol and have a high probability of completing the study.

Exclusion Criteria:

Any one of the following will exclude a subject from being enrolled into the study:

1. Insufficient fluency in English to complete neuropsychological and functional assessments.
2. Concurrent Motor Neuron Disease judged by investigator to have bulbar or upper extremity impairments at baseline that would interfere with neuropsychological assessment, or that are expected to lead to such impairments within one month.
3. Exclusion criteria as listed in Neary criteria. Diagnosis of progressive nonfluent aphasia by Neary criteria.
4. Use of memantine within 4 weeks prior to randomization.
5. Evidence of other neurological or psychiatric disorders which preclude diagnosis of FTD (including, but not limited to, stroke, Parkinson's disease, any psychotic disorder, severe bipolar or unipolar depression, seizure disorder, or head injury with loss of consciousness) within the past year.
6. Concurrent treatment with acetylcholinesterase inhibitors, antipsychotic agents, mood stabilizers (valproate or lithium) or benzodiazepines (other than temazepam or zolpidem), or use of any of these agents within 4 weeks prior to randomization. Atypical antipsychotic agents may be started after the baseline visit if felt to be medically necessary by the investigator and will be recorded as a secondary outcome measure.
7. History of alcohol or substance abuse within 1 year prior to screening, if deemed clinically significant by investigator.
8. Any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
9. Clinically significant lab abnormalities at screening, including Creatinine ≥ 1.7, B12 below laboratory normal reference range or TSH above site's laboratory normal reference range. Subjects with abnormal B12 or TSH levels at screening may be included per investigator's discretion.

9. CT or MRI evidence of any of the following: hydrocephalus, stroke, space-occupying lesion, cerebral infection or any clinically significant CNS disease other than FTD.

10.Systolic blood pressure greater than 180 or less than 90 mm Hg. Diastolic blood pressure greater than 105 or less than 50 mm Hg.

11. Abnormal ECG at screening judged to be clinically significant by the investigator.

12. Use of investigational drugs or participation in investigational drug study within 60 days of screening.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam L. Boxer, M.D., Ph.D., Principal Investigator — University of California, San Francisco; Bruce Miller, M.D., Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - University of California, Los Angeles, Los Angeles, California
  - University California, San Francisco, San Francisco, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland / Case Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Amadoro G, Ciotti MT, Costanzi M, Cestari V, Calissano P, Canu N. NMDA receptor mediates tau-induced neurotoxicity by calpain and ERK/MAPK activation. Proc Natl Acad Sci U S A. 2006 Feb 21;103(8):2892-7. doi: 10.1073/pnas.0511065103. Epub 2006 Feb 13. PMID 16477009
- [Background] Boxer AL, Miller BL. Clinical features of frontotemporal dementia. Alzheimer Dis Assoc Disord. 2005 Oct-Dec;19 Suppl 1:S3-6. doi: 10.1097/01.wad.0000183086.99691.91. PMID 16317256
- [Background] Boxer AL, Trojanowski JQ, Lee VY-M, Miller BL (2005) Frontotemporal Lobar Degeneration. In: Neurodegenerative Diseases: Neurobiology, Pathogenesis and Therapeutics (Beal MF, Lang AE, Ludolph AC, eds), pp 481 - 493. Cambridge, UK: Cambridge University Press.
- [Background] Cullum CM, Saine K, Chan LD, Martin-Cook K, Gray KF, Weiner MF. Performance-Based instrument to assess functional capacity in dementia: The Texas Functional Living Scale. Neuropsychiatry Neuropsychol Behav Neurol. 2001 Apr-Jun;14(2):103-8. PMID 11417663
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Forman MS, Farmer J, Johnson JK, Clark CM, Arnold SE, Coslett HB, Chatterjee A, Hurtig HI, Karlawish JH, Rosen HJ, Van Deerlin V, Lee VM, Miller BL, Trojanowski JQ, Grossman M. Frontotemporal dementia: clinicopathological correlations. Ann Neurol. 2006 Jun;59(6):952-62. doi: 10.1002/ana.20873. PMID 16718704
- [Background] Huey ED, Putnam KT, Grafman J. A systematic review of neurotransmitter deficits and treatments in frontotemporal dementia. Neurology. 2006 Jan 10;66(1):17-22. doi: 10.1212/01.wnl.0000191304.55196.4d. PMID 16401839
- [Background] Josephs KA, Petersen RC, Knopman DS, Boeve BF, Whitwell JL, Duffy JR, Parisi JE, Dickson DW. Clinicopathologic analysis of frontotemporal and corticobasal degenerations and PSP. Neurology. 2006 Jan 10;66(1):41-8. doi: 10.1212/01.wnl.0000191307.69661.c3. PMID 16401843
- [Background] Josephs KA, Duffy JR, Strand EA, Whitwell JL, Layton KF, Parisi JE, Hauser MF, Witte RJ, Boeve BF, Knopman DS, Dickson DW, Jack CR Jr, Petersen RC. Clinicopathological and imaging correlates of progressive aphasia and apraxia of speech. Brain. 2006 Jun;129(Pt 6):1385-98. doi: 10.1093/brain/awl078. Epub 2006 Apr 13. PMID 16613895
- [Background] Kertesz A, Davidson W, Fox H. Frontal behavioral inventory: diagnostic criteria for frontal lobe dementia. Can J Neurol Sci. 1997 Feb;24(1):29-36. doi: 10.1017/s0317167100021053. PMID 9043744
- [Background] Kertesz A, McMonagle P, Blair M, Davidson W, Munoz DG. The evolution and pathology of frontotemporal dementia. Brain. 2005 Sep;128(Pt 9):1996-2005. doi: 10.1093/brain/awh598. Epub 2005 Jul 20. PMID 16033782
- [Background] Lipton SA. Paradigm shift in neuroprotection by NMDA receptor blockade: memantine and beyond. Nat Rev Drug Discov. 2006 Feb;5(2):160-70. doi: 10.1038/nrd1958. PMID 16424917
- [Background] Lipton SA, Rosenberg PA. Excitatory amino acids as a final common pathway for neurologic disorders. N Engl J Med. 1994 Mar 3;330(9):613-22. doi: 10.1056/NEJM199403033300907. No abstract available. PMID 7905600
- [Background] Mendez MF, Shapira JS, McMurtray A, Licht E. Preliminary findings: behavioral worsening on donepezil in patients with frontotemporal dementia. Am J Geriatr Psychiatry. 2007 Jan;15(1):84-7. doi: 10.1097/01.JGP.0000231744.69631.33. PMID 17194818
- [Background] Moretti R, Torre P, Antonello RM, Cattaruzza T, Cazzato G, Bava A. Rivastigmine in frontotemporal dementia: an open-label study. Drugs Aging. 2004;21(14):931-7. doi: 10.2165/00002512-200421140-00003. PMID 15554751
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Neary D, Snowden JS, Gustafson L, Passant U, Stuss D, Black S, Freedman M, Kertesz A, Robert PH, Albert M, Boone K, Miller BL, Cummings J, Benson DF. Frontotemporal lobar degeneration: a consensus on clinical diagnostic criteria. Neurology. 1998 Dec;51(6):1546-54. doi: 10.1212/wnl.51.6.1546. PMID 9855500
- [Background] Orgogozo JM, Rigaud AS, Stoffler A, Mobius HJ, Forette F. Efficacy and safety of memantine in patients with mild to moderate vascular dementia: a randomized, placebo-controlled trial (MMM 300). Stroke. 2002 Jul;33(7):1834-9. doi: 10.1161/01.str.0000020094.08790.49. PMID 12105362
- [Background] Pijnenburg YA, Sampson EL, Harvey RJ, Fox NC, Rossor MN. Vulnerability to neuroleptic side effects in frontotemporal lobar degeneration. Int J Geriatr Psychiatry. 2003 Jan;18(1):67-72. doi: 10.1002/gps.774. PMID 12497558
- [Background] Reisberg B, Doody R, Stoffler A, Schmitt F, Ferris S, Mobius HJ; Memantine Study Group. Memantine in moderate-to-severe Alzheimer's disease. N Engl J Med. 2003 Apr 3;348(14):1333-41. doi: 10.1056/NEJMoa013128. PMID 12672860
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Royall DR, Mahurin RK, Gray KF. Bedside assessment of executive cognitive impairment: the executive interview. J Am Geriatr Soc. 1992 Dec;40(12):1221-6. doi: 10.1111/j.1532-5415.1992.tb03646.x. PMID 1447438
- [Background] Tariot PN, Farlow MR, Grossberg GT, Graham SM, McDonald S, Gergel I; Memantine Study Group. Memantine treatment in patients with moderate to severe Alzheimer disease already receiving donepezil: a randomized controlled trial. JAMA. 2004 Jan 21;291(3):317-24. doi: 10.1001/jama.291.3.317. PMID 14734594
- [Background] Wilcock G, Mobius HJ, Stoffler A; MMM 500 group. A double-blind, placebo-controlled multicentre study of memantine in mild to moderate vascular dementia (MMM500). Int Clin Psychopharmacol. 2002 Nov;17(6):297-305. doi: 10.1097/00004850-200211000-00005. PMID 12409683
- [Background] Winblad B, Poritis N. Memantine in severe dementia: results of the 9M-Best Study (Benefit and efficacy in severely demented patients during treatment with memantine). Int J Geriatr Psychiatry. 1999 Feb;14(2):135-46. doi: 10.1002/(sici)1099-1166(199902)14:23.0.co;2-0. PMID 10885864
- [Result] Boxer AL, Knopman DS, Kaufer DI, Grossman M, Onyike C, Graf-Radford N, Mendez M, Kerwin D, Lerner A, Wu CK, Koestler M, Shapira J, Sullivan K, Klepac K, Lipowski K, Ullah J, Fields S, Kramer JH, Merrilees J, Neuhaus J, Mesulam MM, Miller BL. Memantine in patients with frontotemporal lobar degeneration: a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2013 Feb;12(2):149-56. doi: 10.1016/S1474-4422(12)70320-4. Epub 2013 Jan 2. PMID 23290598
- See also: UCSF Memory and Aging Center — http://memory.ucsf.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients from nine US academic dementia research centres with expertise in the diagnosis of FTD. Study visits occurred between December 12, 2007, and May 7, 2012.
Pre-assignment Details: 100 subjects were assessed for eligibility. 19 were excluded prior to randomization. 81 were randomized. 16 subjects did not meet inclusion criteria and 3 declined to participate.
Groups:
- Memantine: Memantine 10mg administered orally twice daily
- Placebo: Placebo (inactive tablets identical to memantine 10mg tablets)
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 39 (subjects randomized to memantine cohort) | 42 (subjects randomized to placebo cohort)
Completed | 37 (subjects completed 26 weeks treatment in memantine cohort) | 39 (subjects completed 26 weeks treatment in placebo cohort)
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 25 | 43
  >=65 years | 21 | 17 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (2.8) | 66.2 (2.3) | 66.0 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 19 | 32 | 51
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropsychiatric Inventory (NPI)
Description: NPI:12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, nighttime behavior. A screening question is asked about each sub-domain. If the responses to these questions indicate that the patient has problems with a particular sub-domain of behavior, the caregiver is only then asked all the questions about that domain, rating the frequency of the symptoms on a 4-point scale, their severity on a 3-point scale, and the distress the symptom causes them on a 5-point scale. Severity(1=Mild to 3=Severe),frequency(1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score(range 0-12). Total score=sum of each domain score(range 0-144);higher score=greater behavioral disturbances;negative change score from baseline=improvement.
Time Frame: Baseline, 26 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 37 | 39
units on a scale | -1.9 [-6.1 to 2.3] | 0.3 [-4 to 4.7]

2. Primary Outcome: Clinical Global Impression of Change (CGIC)
Description: The scale is rated on a 7-point scale, using a range of responses from 1 (very much improved) through 7 (very much worse). The clinician compares the participant's current condition to the condition at admission to the project.
Time Frame: 26 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 37 | 39
units on a scale | 4.4 [3.7 to 5.2] | 4.8 [4.8 to 5.1]

3. Secondary Outcome: Longitudinal Changes From Baseline to 26 Weeks for Test Battery: CDR-SB, FAQ, TFLS, MMSE, EXIT25, UPDRS, Boston Naming Test
Description: Clinical dementia rating sum of boxes CDR-SB (0-18) high scores indicate high impairment.
  Functional activities questionnaire FAQ (0-30) high scores indicate high impairment.
  Texas functional living scale TFLS (0 to 52) high scores suggest better instrumental activities of daily living functioning.
  Mini-Mental State Examination MMSE (0-30) low scores indicate low cognition. The executive interview EXIT25 (0 to 50) high scores indicate more executive impairment.
  A modified unified Parkinson's disease rating scale UPDRS (0-199) high scores indicate worse disability.
  Boston naming test (0-15) low scores indicate more retrieval difficulties.
Time Frame: Baseline and 26 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 37 | 39
units on a scale
  CDR-SB | 1.5 [0.9 to 2.1] | 1.5 [0.8 to 2.1]
  FAQ | 4.3 [2.7 to 6.0] | 2.9 [1.0 to 4.7]
  TFLS | -3.7 [-5.7 to -1.7] | -2.8 [-4.4 to -1.1]
  MMSE | -1.2 [-2.5 to 0.1] | -0.9 [-1.8 to 0.0]
  EXIT25 | 1.9 [-0.1 to 3.9] | 0.7 [-1.1 to 2.4]
  UPDRS | 1.7 [-0.1 to 3.4] | 1.4 [-0.7 to 3.4]
  Boston naming test | -1.4 [-2.9 to 0.0] | 0.7 [0.3 to 1.2]

4. Secondary Outcome: Longitudinal Changes From Baseline to 26 Weeks for Test Battery: Letter Fluency, Category Fluency, Digit Symbol, Digits Backwards
Description: Letter fluency, score is number of words recalled starting with a specified letter for 60 seconds. There are 3 trials, with 3 different letters. The total number of correct responses is totaled for all 3 trials for the score. Low scores indicate high impairment
  Category fluency, score is number of items generated belonging to a specific category (such as animals) in 60 seconds, low scores indicate high impairment.
  Digit symbol, score is number of symbols that correctly corresponded to the random numerals entered in the form in 90 seconds. Participants are given a table of numerals with matching symbols, and a form with random numerals with open spaces. Low scores indicate high impairment.
  Digits backwards, score is number of digits backwards recalled (range: 0-14), The participant hears a list of digits and is asked to repeat the digits backwards. Low scores indicate high impairment.
Time Frame: Baseline and 26 Weeks
Measure: Mean (95% Confidence Interval); unit: number of items recalled
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 37 | 39
number of items recalled
  Letter fluency | -0.1 [-1.2 to 1.1] | -0.3 [-1.1 to 0.4]
  Category fluency | -0.5 [-1.9 to 0.9] | -0.7 [-2.7 to 1.3]
  Digit symbol | -3.9 [-7.5 to -0.3] | 4.2 [1.7 to 10.1]
  Digits backwards | 0.1 [-0.3 to 0.5] | -0.2 [-0.5 to 0.2]

5. Secondary Outcome: Number of Participants Starting Antipsychotic Therapy
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 37 | 39
Participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/39 | 2/42
Other Adverse Events (participants affected / at risk) | 28/39 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=39) | Placebo (N=42)
diverticulitis leading to hospital admission (Gastrointestinal disorders) | 0 | 1
vasovagal episode (Nervous system disorders) | 0 | 1
right-sided facial weakness and loss of consciousness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=39) | Placebo (N=42)
fatigue (General disorders) | 1 | 1
language problems (Psychiatric disorders) | 3 | 0
memory loss (Psychiatric disorders) | 2 | 0
diverticulitis (Gastrointestinal disorders) | 0 | 2
nausea (Gastrointestinal disorders) | 0 | 3
abrasion (Injury, poisoning and procedural complications) | 2 | 0
fall (Injury, poisoning and procedural complications) | 5 | 2
dizziness (Nervous system disorders) | 2 | 2
headache (Nervous system disorders) | 1 | 3
agitation (Nervous system disorders) | 0 | 2
back pain (Nervous system disorders) | 2 | 0
behavioral rigidity (Psychiatric disorders) | 1 | 1
inappropriate sexual behavior (Psychiatric disorders) | 0 | 4
insomnia (Psychiatric disorders) | 0 | 4
obsessive compulsive symptoms (Psychiatric disorders) | 2 | 1
somnolence (Psychiatric disorders) | 1 | 1
urinary tract infection (Renal and urinary disorders) | 2 | 0
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
urinary frequency (Renal and urinary disorders) | 1 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Lower enrollment than planned may have limited ability detect a treatment effect; Small size of semantic dementia group limits generalizability of results to FTD syndrome; Newer tools have been developed to better capture FTD-specific behaviors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No